CLINICAL TRIAL: NCT02850874
Title: Hyperthermic Intraperitoneal Chemotherapy as Neoadjuvant Treatment for Resectable Pancreatic Adenocarcinoma: A Prospective, Phase II, Proof-of-concept Study
Brief Title: HIPEC as Neoadjuvant Treatment for Resectable Pancreatic Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual rate
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-16-05A
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Neoplasms; Pancreatic Adenocarcinoma
Keywords: hyperthermic intraperitoneal chemotherapy; perioperative systemic chemotherapy; peritoneal disease
MeSH Terms: conditions — Pancreatic Neoplasms; Peritoneal Diseases | interventions — Hyperthermic Intraperitoneal Chemotherapy; Pancreaticoduodenectomy; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIPEC (Experimental): Immediately following laparoscopy for diagnosis and staging of disease, closed neoadjuvant hyperthermic intraperitoneal chemotherapy (HIPEC) will be performed using the anatomical site of the laparoscopic procedure in the same operative encounter. Perfusion will be initiated with 4-6 L of 1.5% dextrose at a 500 mL/min flow rate with manual agitation of the abdominal wall. Once the temperature in the abdomen becomes stable above 40°C, perfusate volume will be reduced to 1.5 L/m sq, and gemcitabine (GEMZAR®) will be instilled into the abdomen (1000 mg/m sq) for 90 min. Neoadjuvant chemotherapy with gemcitabine will be administered prior to open pancreaticoduodenectomy by the standard Whipple or pylorus-preserving approach. Adjuvant systemic chemotherapy with gemcitabine will be administered for 6 months (including period of neoadjuvant therapy) according to established institutional protocol.
  Interventions: Procedure: Hyperthermic intraperitoneal chemotherapy; Procedure: Open pancreaticoduodenectomy; Drug: Gemcitabine
- Historical Control (Other): Case-matched historical controls will have received neoadjuvant chemotherapy with gemcitabine prior to open pancreaticoduodenectomy (PD) by the standard Whipple or pylorus-preserving approach. Adjuvant systemic chemotherapy (SCT) with gemcitabine will be administered for 6 mo (including period of neoadjuvant therapy) according to established institutional protocol.
  Interventions: Procedure: Open pancreaticoduodenectomy; Drug: Gemcitabine

INTERVENTIONS:
Procedure: Hyperthermic intraperitoneal chemotherapy — HIPEC in this study involves the washing of the peritoneal cavity with a heated (40-48°C), (1000 mg/m sq) solution of gemcitabine in 1.5% dextrose for 90 min. Compared with systemic delivery of chemotherapy, intraperitoneal delivery can increase site-specific concentration of chemotherapeutic agents and decrease duration of perfusion, vascular complications, and systemic toxicity. The use of heated chemotherapeutic agents, compared to conventional protocols, has been shown to increase direct cytotoxicity to malignant cells and augment penetration into tumors.
  Other Names: HIPEC
  Arms: HIPEC
Procedure: Open pancreaticoduodenectomy — Tumors of the pancreatic head will be surgically removed by open PD (standard and pylorus-preserving approaches) with the aim of achieving en bloc R0 tumor resection (no macroscopic residual cancer remaining). In all patients, a lymphadenectomy will be performed along the hepatoduodenal ligament, common hepatic artery, vena cava, and the interaortocaval and right side of the superior mesenteric artery. In cases with portal vein involvement, a venous resection will be performed to achieve R0 resection. Patients with arterial infiltration by the tumor will be deemed locally nonresectable and will be excluded from analysis.
  Established, routine surgical and ERAS protocols will be followed for pre-, intra-, and postoperative care of patients. Patients will be discharged after postoperative day 5 if tolerating oral intake and showing no signs or symptoms of complications.
  Other Names: Whipple procedure; Pylorus-preserving pancreaticoduodenectomy (PPPD)
Drug: Gemcitabine — Neoadjuvant and adjuvant systemic chemotherapy will be administered to all PDAC patients with the aim of diminishing the tumor burden and maximizing the chance of complete surgical resection. Gemcitabine (GEMZAR®) will be administered for 6 months (including period of neoadjuvant therapy) according to established institutional guidelines for dosing, frequency, duration, administration route, and setting.
  Other Names: GEMZAR®

SUMMARY:
This single-center, prospective proof-of-concept study is designed to evaluate the surgical outcomes and clinicopathologic results of neoadjuvant hyperthermic intraperitoneal chemotherapy (HIPEC) in conjunction with perioperative systemic chemotherapy (SCT; neoadjuvant and adjuvant) and pancreaticoduodenectomy (PD) in a small cohort of patients having T1-T3 resectable pancreatic ductal adenocarcinoma (PDAC) with one or more high-risk clinical features. The investigators hypothesize that HIPEC administered in this clinical course will reduce postoperative peritoneal disease recurrence. The investigators also expect that local recurrence of disease will be reduced. The primary aim of this study is to compare 2-year peritoneal disease-free survival between patients receiving the experimental therapy (neoadjuvant HIPEC + SCT + PD) with historical controls receiving standard therapy (SCT + PD). Secondary aims are to determine the clinical feasibility and outcomes of neoadjuvant HIPEC for resectable PDAC using patient demographics and disease characteristic data.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of pancreatic ductal adenocarcinoma (PDAC) confined to the head of the pancreas classified as T1-T3 with one or more of the following high-risk clinical features:

  * Carbohydrate antigen (CA) 19-9 greater than 1,000 U/mL with a normal bilirubin;
  * Vascular involvement; and/or
  * Suspicious regional lymphadenopathy
* Intention to undergo open pancreaticoduodenectomy (standard Whipple or pylorus-preserving pancreaticoduodenectomy) as treatment for PDAC
* Adequate clinical condition to undergo preoperative (neoadjuvant) hyperthermic intraperitoneal chemotherapy
* Adequate clinical condition to undergo perioperative systemic chemotherapy
* White blood cell count of at least 3000/mL
* Platelet count of at least 100,000/mL
* Normal creatinine (< 2 mg/dL) or creatinine clearance of at least 50 mL/min
* Willing and able to give informed consent

Exclusion Criteria:

* Evidence of locoregional spread (carcinomatosis of peritoneal surfaces, mesenteric arteries, or body/tail of pancreas) or distant (liver, lung, or other) metastases (histological, CT, or MRI confirmation)
* Non-curative intent of treatment (≥R2 resection)
* Body mass index (BMI) > 35
* Previous history of pancreatic resections for tumors in the body and/or tail of the pancreas, distal cholangiocarcinoma, duodenal carcinoma, neuroendocrine tumors, cyst-adenocarcinoma, or solid and papillary tumors.
* Unstable or uncompensated respiratory or cardiac disease
* Severe hepatic or renal dysfunction
* Bleeding diathesis or coagulopathy
* Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Peritoneal disease-free survival | 2 years
  Peritoneal disease-free survival is defined as the time between staging laparoscopy confirming no peritoneal disease (at the time of HIPEC treatment) and regional recurrence of pancreatic ductal adenocarcinoma on the peritoneal surfaces as determined by diagnostic imaging. This definition is exclusive of recurrence status in the pancreatic remnant after resection.

SECONDARY OUTCOMES:
Overall survival | 1, 2, 3, 5 years
Local disease-free survival | 2 years
  Local disease-free survival is defined as the time between staging laparoscopy (at the time of HIPEC treatment) and local recurrence of pancreatic ductal adenocarcinoma in the pancreatic remnant as determined by diagnostic imaging.
Postoperative morbidity | 1 and 3 months
Postoperative mortality | 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dionisios Vrochides, MD PhD FACS, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided